CLINICAL TRIAL: NCT06382597
Title: Four Weeks of Nordic Hamstring Exercises Impact the Strength and Balance of the Hamstring Muscle Group
Status: Completed | Type: Observational
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Other Study IDs: AWFiS/2024_2_P-GM
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Hamstring Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nordic Hamstring Exercise: The subjects will be randomly divided into two research groups. The first research group will undergo a 4-week Nordic Hamstring Exercise training, the second research group will be a control group performing traditional exercises.
  Interventions: Other: Nordic hamstring exercise

INTERVENTIONS:
Other: Nordic hamstring exercise — Nordic Hamstring Exercise involves a controlled descent of the upright torso from a vertical kneeling position forward towards the ground (parallel to the ground) and returning to the starting position. The ankle joints are stabilized by the other person's grip during a series of exercises.

SUMMARY:
The aim of the study is to assess the impact of 4 weeks of eccentric Nordic Hamstring Exercise training on changes in the hamstring muscle group, as well as to analyze parameters such as maximum muscle strength of the knee flexors, RFD (rate of force development) and static balance, dynamics for the dominant leg.

DETAILED DESCRIPTION:
Research procedure: Nordic Hamstring Exercise training covers a period of 4 weeks, during which the volunteer exercises 3 times a week for 3 sets, each set consisting of 3 repetitions of NHE. Before starting eccentric exercises, you will warm up for 15 minutes. After each series, there will be a 2-minute passive break, during which the subject will rest. In the first week, the subject will exercise under the supervision of the instructor, in the next three weeks the subject will exercise at home after prior instruction.

ELIGIBILITY:
Inclusion Criteria:

* healthy people aged 19-26,
* no injuries,
* athletes, people practicing sports as amateurs

Exclusion Criteria:

* during the period of greatest training load related to the discipline,
* overload changes in the joints: knee, hip and lumbar-sacral,
* pain,
* muscle fatigue, overtraining,
* in strength sports a few weeks before the start,
* inflammation of the osteoarticular and ligamentous elements of the lower limbs,
* previous injuries, surgical procedures within 6 months before the intervention

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will involve students of the Academy of Physical Education and Sport in Gdańsk, aged 19-26 who practice amateur football.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Biodex Balance System | 15 min
  The medial-lateral stability index (MLSI), anteroposterior stability index (APSI) and general static and dynamic stability index will be assessed for both limbs and the dominant leg

SECONDARY OUTCOMES:
Biodex System | 20 min
  The maximum muscle strength of the hamstring group will be assessed for both legs

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Podczarska-Głowacka, Study Chair — Department of Basic Physiotherapy, Gdansk University of Physical Education and Sport, Gdansk, Poland
Locations (1):
- Academy of Physical Education in Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No